CLINICAL TRIAL: NCT00072007
Title: 2-CDA and Rituximab as Remission Induction and Rituximab as In Vivo Purging Prior to Peripheral Stem Cell Mobilization in Patients With Chronic Lymphocytic Leukemia (CLL) - A Prospective Multicenter Phase II Trial
Brief Title: Cladribine and Rituximab as Remission Induction Therapy Followed By Rituximab and Stem Cell Mobilization in Treating Patients With CLL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 34/02; EU-20321
Record Dates: First submitted 2003-11-04; First posted 2003-11-06 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Leukemia
Keywords: B-cell chronic lymphocytic leukemia; refractory chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Filgrastim; Rituximab; VAP-cyclo protocol; Cladribine; Cyclophosphamide; Doxorubicin; Prednisone; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: filgrastim — filgrastim
Biological: rituximab — rituximab
Drug: CHOP regimen — CHOP regimen
Drug: cladribine — cladribine
Drug: cyclophosphamide — cyclophosphamide
Drug: doxorubicin hydrochloride — doxorubicin hydrochloride
Drug: prednisone — prednisone
Drug: vincristine sulfate — vincristine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cladribine, use different ways to stop cancer cells from dividing so they stop growing or die. Monoclonal antibodies, such as rituximab, can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Combining cladribine with rituximab may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving cladribine and rituximab as remission induction therapy together with rituximab and stem cell mobilization in treating patients with chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy and tolerability of cladribine and rituximab as remission induction therapy in patients with chronic lymphocytic leukemia.
* Determine the complete remission rate in patients treated with this regimen.

Secondary

* Determine the very good partial remission rate and nodular partial remission rate in patients treated with this regimen.
* Determine the toxicity of this regimen, in terms of hemotoxicity and infection rate, in these patients.
* Determine the efficacy of in vivo purging with rituximab measured by immunophenotyping in these patients.
* Determine the feasibility of stem cell harvest in these patients after treatment with this induction therapy regimen and in vivo purging with rituximab.

OUTLINE: This is a multicenter study.

* Remission induction: Patients receive cladribine subcutaneously (SC) on days 1-5. During courses 2-4, patients also receive rituximab IV on day 1. Treatment repeats every 28 days for up to 4 courses in the absence of unacceptable toxicity. If unacceptable toxicity persists, patients receive rituximab alone.

Patients not achieving a complete remission (CR), very good partial remission (VGPR), or nodular partial remission (NPR) receive CHOP chemotherapy comprising cyclophosphamide IV, doxorubicin IV, and vincristine IV on day 1 and oral prednisone on days 1-5. Treatment repeats every 21 days for up to 4 courses or until patients achieve a CR, VGPR, or NPR.

Patients achieving a CR, VGPR, or NPR proceed to stem cell mobilization and in vivo purging.

* Stem cell mobilization and in vivo purging: Beginning 8-10 weeks after the first day of the last course of remission induction or CHOP, patients receive rituximab IV on days 1 and 8, cyclophosphamide IV over 4 hours on day 2, and filgrastim (G-CSF) SC daily beginning on day 4 and continuing until the last day of apheresis. Patients undergo apheresis on days 11-14.

PROJECTED ACCRUAL: A total of 17-41 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of B-cell chronic lymphocytic leukemia (CLL)

  * CD5 positive and CD23 positive
  * Binet stage B, C, or progressive A
* Newly diagnosed disease OR no more than 1 prior alkylating agent regimen (e.g., chlorambucil or cyclophosphamide with or without prednisone)

PATIENT CHARACTERISTICS:

Age

* 18 to 65

Performance status

* WHO 0-2

Life expectancy

* Not specified

Hematopoietic

* No autoimmune hemolytic anemia
* No immune thrombocytopenia

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* Alkaline phosphatase no greater than 2.5 times ULN*
* AST and ALT no greater than 2.5 times ULN* NOTE: *Unless clearly related to CLL liver involvement

Renal

* Creatinine clearance greater than 50 mL/min

Cardiovascular

* Ejection fraction at least 50%
* No severe heart failure
* No unstable angina pectoris
* No significant arrhythmia requiring chronic treatment
* No myocardial infarction within the past 3 months

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 12 months after study participation
* HIV negative
* No active infection
* No positive Coombs' test
* No history of significant neurologic or psychiatric disorders, including psychotic disorders or dementia
* No seizure disorder
* No other malignancy within the past 5 years except nonmelanoma skin cancer or adequately treated carcinoma in situ of the cervix
* No prior allergic reaction or hypersensitivity to study drugs or attributed to compounds of similar chemical or biological composition to study drugs or other study agents
* No uncontrolled diabetes mellitus
* No gastric ulcers
* No active autoimmune disease
* No alcohol or drug abuse
* No other concurrent serious underlying medical condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* No prior purine analogs (e.g., cladribine or fludarabine)

Endocrine therapy

* Not specified

Radiotherapy

* No concurrent radiotherapy

Surgery

* Not specified

Other

* More than 30 days since prior clinical trial participation
* No other concurrent experimental drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2002-06; Primary Completion 2003-03 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Complete-remission rate after induction | 30 days

SECONDARY OUTCOMES:
Very good partial remission and nodular partial remission after induction | 30 days
Toxicity (hematotoxicity and infection rate) at 30 days following study treatment | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Reinhard Zenhaeusern, MD, Study Chair — Insel Gruppe AG, University Hospital Bern
Locations (11):
- Switzerland (11):
  - Kantonspital Aarau, Aarau
  - Oncology Institute of Southern Switzerland, Bellinzona
  - Inselspital Bern, Bern
  - Spitaeler Chur AG, Chur
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - Kantonsspital, Luzerne, Luzerne
  - Hopital des Cadolles, Neuchatel, Neuchâtel
  - Praxis Dr. Beretta, Rheinfelden
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Onkozentrum, Zurich
  - UniversitaetsSpital Zuerich, Zurich

REFERENCES:
- [Result] Leupin N, Schuller JC, Solenthaler M, Heim D, Rovo A, Beretta K, Gregor M, Bargetzi MJ, Brauchli P, Himmelmann A, Hanselmann S, Zenhausern R. Efficacy of rituximab and cladribine in patients with chronic lymphocytic leukemia and feasibility of stem cell mobilization: a prospective multicenter phase II trial (protocol SAKK 34/02). Leuk Lymphoma. 2010 Apr;51(4):613-9. doi: 10.3109/10428191003624231. PMID 20218808
- [Result] Leupin N, Schuller JC, Solenthaler M, et al.: The combination of 2-CDA and rituximab in patients with chronic lymphocytic leukemia (CLL): a prospective multicenter phase II trial (SAKK 34/02). [Abstract] Blood 110 (11): A-2057, 2007.